CLINICAL TRIAL: NCT00146549
Title: A Randomized Phase III Study of Trastuzumab (Herceptin) in Combination With Either Vinorelbine (Navelbine), or Taxane-based Chemotherapy in Patients With HER2 Overexpressing Metastatic Breast Cancer
Brief Title: Trastuzumab in Combination With Vinorelbine or Taxane-Based Chemotherapy in Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Massachusetts General Hospital (Other); Brigham and Women's Hospital (Other); North Shore Medical Center (Other); GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01-087
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2009-11-02 (Estimated); Status verified 2009-10

CONDITIONS: Breast Cancer; Stage IV Breast Cancer
Keywords: HER2-positive Breast cancer; HER2 overexpressing; trastuzumab; Herceptin; vinorelbine; Navelbine; Taxotere; taxol
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Vinorelbine; Paclitaxel; Docetaxel

INTERVENTIONS:
Drug: Trastuzumab
Drug: Vinorelbine
Drug: Paclitaxel
Drug: Docetaxel

SUMMARY:
The purpose of this study is to compare two different combinations of chemotherapy with trastuzumab as initial treatment for HER2 positive advanced breast cancer. Half of the patients will receive trastuzumab in combination with a taxane form of chemotherapy (either paclitaxel or docetaxel), while the other group will receive trastuzumab in combination with vinorelbine.

DETAILED DESCRIPTION:
* All patients will receive trastuzumab then be randomized into one of two arms. Arm A: Trastuzumab in combination with weekly vinorelbine and Arm B: Trastuzumab in combination with a weekly taxane-based regimen, either paclitaxel or docetaxel, chosen at the discretion of the investigator.
* Treatment is administered on an outpatient basis. Trastuzumab is administered weekly. There is a one-time loading dose for the first week of the first cycle. For that initial treatment, only, the trastuzumab dose is 4mg/kg. The dose for all subsequent weekly trastuzumab treatments is 2mg/kg.
* Arm A: vinorelbine is administered every week and the dose is adjusted based on the absolute neutrophil count for that week. Vinorelbine is given after trastuzumab.
* Arm B: Either paclitaxel given weekly (dose bases on absolute neutrophil count) or docetaxel given on weeks 1,2,3,5,6,7 of each 8-week cycle (dose based upon absolute neutrophil count). Patients on paclitaxel will also receive dexamethasone, diphenhydramine and ranitidine to help prevent allergic or hypersensitivity reactions. Patients on docetaxel will receive dexamethasone to help reduce fluid retention or edema.
* Every 8 weeks the patients cancer will be re-evaluated to see if the treatment is working. If the treatment appears to be working, treatment will continue. Standard radiological testing (x-rays, CT scan, radioactive drug scans, or MRI's) will be used to follow the disease treatment.
* Heart function will be measured after 16 weeks to be sure it is safe to continue treatment.
* Every 8 weeks, patients' will be asked to complete a brief written survey that asks about symptoms and side effects.
* Patients' will remain on the treatment as long as there is no disease progression or unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed invasive breast cancer, with stage IV disease
* Tumors must be HER2 overexpressing
* Measurable disease, defined as a least one lesion that can be accurately measured in at least one dimension
* 18 years of age or older
* Life expectancy of greater than 6 months
* ECOG performance status of 0-2
* ANC count > 1,500/mm3
* Platelets > 100,000/mm3
* Total bilirubin < 1.5 mg/dl
* AST/ALT < 115 U/I
* Creatinine < 2.0 mg/dl
* Glucose < 200 mg/dl
* LVEF > 50%

Exclusion Criteria:

* Prior chemotherapy or prior trastuzumab therapy for metastatic breast cancer
* Concurrent hormonal therapy, chemotherapy, or radiation treatments
* Pregnant or lactating women
* Known brain metastases or leptomeningeal carcinomatosis
* History of grade 3 or 4 allergic reactions attributed to compounds of similar chemical or biologic composition to the agents in this study
* Pre-existing neuropathy from any cause in excess of grade 1
* Uncontrolled intercurrent illness
* History of other non-breast cancer malignancy except for carcinoma in situ of the cervix or non-melanoma skin cancer
* Patients taking macrolide antibiotics, ketoconazole, or AZT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2001-08; Primary Completion 2007-08 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To compare the overall response rate for patients receiving trastuzumab in combination with either vinorelbine or taxane-based chemotherapy.

SECONDARY OUTCOMES:
Characterization of the time to disease progression and time to treatment failure for patients receiving trastuzumab with either vinorelbine or taxane-based chemotherapy
Characterization of side effects for both treatments
analysis of quality of life for patients receiving either treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Harold Burstein, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts